CLINICAL TRIAL: NCT05055882
Title: Auvergne-Rhône-Alpes-Limousin Research Database for Still's Diseases in Children and Adults
Acronym: AURAL-STILL
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2021_003
Record Dates: First submitted 2021-09-08; First posted 2021-09-24 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Still Disease
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children and adult diagnosed with Still's disease in Auvergne-Rhône-Alpes-Limousin hospital: children and adult with Still's disease in Auvergne-Rhône-Alpes-Limousin hospital
  Interventions: Other: children and adult with Still's disease in Auvergne-Rhône-Alpes-Limousin hospital

INTERVENTIONS:
Other: children and adult with Still's disease in Auvergne-Rhône-Alpes-Limousin hospital — Comparison of Adult-Onset Still's disease phenotypes

SUMMARY:
Adult-Onset Still's disease is a polygenic autoinflammatory disease of unknown etiology. The autoinflammatory character individualizes it from autoimmune autoantibody diseases. Clinically, it results in the classic triad associating hectic fever, evanescent rash and arthritis. Although it is benign in the vast majority of cases, life-threatening complications can occur. By definition, the disease affects adults over 16 years of age, however most experts now agree that the adult form and the pediatric form belong to a pathological continuum: Still's disease. In the absence of a specific biomarker, the diagnosis is still based on clinical and biological criteria, after the exclusion of differential diagnoses.

Classically, three evolutionary profiles of Adult-Onset Still's disease are individualized, depending on the evolution of symptoms over time:

* a monocyclic systemic form (30% of cases) characterized by clear systemic symptoms and in the foreground compared to the articular signs. This form evolves over several weeks to several months (on average 9 months), without exceeding a year. By definition, there is no recurrence;
* a polycyclic systemic form (30% of cases) defined by the occurrence of at least two systemic or joint episodes, separated by clinical remission intervals greater than two months, or even several years. The symptoms of relapses are not always the same as the initial symptoms. The number and severity of relapses is unpredictable and varies widely from patient to patient, but symptoms tend to become less severe over time.
* a chronic form, with predominant joint involvement (40%), resembling seronegative rheumatoid arthritis. Systemic signs are present during the first outbreaks of the disease. Subsequently, rheumatoid arthritis evolves on its own and one can see joint destruction or conversely ankylosing developments such as the classic bilateral, non-erosive fusing carpitis.

There are reasons to believe that the evolving profile of patients has changed since the emergence and generalization of biotherapies. Furthermore, no prognostic factor for the progression of Adult-Onset Still's disease has been found so far. The differences between pediatric and adult forms need to be confirmed and becoming pediatric forms in adulthood is poorly described.

The objective of this study is to set up a regional research database (Auvergne-Rhône-Alpes-Limousin) in order to describe the characteristics, treatment and evolution of patients with Still's disease.

ELIGIBILITY:
Inclusion Criteria:

* children and adult diagnosed with Still's disease in Auvergne-Rhône-Alpes-Limousin hospital

Exclusion Criteria:

* Not applicable

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children and adult diagnosed with Still's disease in Auvergne-Rhône-Alpes-Limousin hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
validation of classification criteria | at inclusion
  number of participants with clinical and biological abnormalities, as assessed in the Yamaguchi and Fautrel criteria

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Hôpital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier de Valence, Valence, Drome
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospitalier de Bourg en Bresse, Bourg-en-Bresse
  - Centre Hospitalier Bourgoin Jallieu, Bourgoin
  - Centre Hospitalier de Chambéry, Chambéry
  - Centre Hospitalier de Châlon sur Saône, Châlon Sur Saône
  - Centre Hospitalier Alpes-Léman (CHAL), Contamine-sur-Arve
  - Centre Hospitalier du puy en velay, Le Puy-en-Velay
  - Centre Hospitalier de Limoges, Limoges
  - Hopital Saint Luc Saint Joseph, Lyon
  - Hospices Civils de Lyon - Edouard Herriot, Lyon
  - Centre Hospitalier de Montélimar, Montélimar
  - Centre Hospitalier Vienne, Vienne
  - Centre Hospitalier de Villefranche, Villefranche-sur-Saône
  - Médipôle de Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared